CLINICAL TRIAL: NCT03420027
Title: Evaluation of the Feasibility of the MACOCHA Score and Indication of Endotracheal Intubation in Prehospital and Emergency Room: a Prospective Observational Study
Brief Title: Prehospital and Emergency Feasibility of MACOCHA Score Assessment to Predict Difficult Tracheal Intubation
Acronym: E-MAC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2017- 14; 2017-A02885-48 (IDRCB number) (Other: French Ministry of Health)
Record Dates: First submitted 2018-01-28; First posted 2018-02-05 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Intubation, Intratracheal; Emergency Medicine
Keywords: predictive score; difficult intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire to be filled in by investigators — A simple seven-item questionnaire will be filled in by the investigator before performing urgent tracheal intubation. This intubation, which will be performed as done in routine care, does not constitute a study specific intervention

SUMMARY:
A seven-item simplified score (the MACOCHA score) has been validated to predict difficult tracheal intubation in intensive care unit patients. In the prehospital or in the emergency department settings, no such validated predictive score is available yet. The aim of the present study is to assess the feasibility the quick calculation of the MACOCHA score before emergent intubation, in the prehospital and emergency department contexts.

DETAILED DESCRIPTION:
All patients who will have to undergo emergent tracheal intubation for any reason in the prehospital context or at the emergency department at a single 1100-bed regional and teaching hospital in France, will be included in this observational, prospective study, provided that neither the patient him/herself, if capable, or next-of-kin if present have declined participation.

Items of the MACOCHA score will be recorded before intubation by investigators, who are all certified emergency physicians skilled with urgent tracheal intubation.

For any intubation procedure, either in the out-of-hospital context or in the Emergency Department, one of these emergency physicians is always present.

The feasibility the quick MACOCHA score calculation before urgent intubation will be assessed by the number and percentages of patients for whom all the seven items of the score have been collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 yrs
* Patient who have to undergo rapid sequence tracheal intubation as judged by the Emergency Physician

Exclusion Criteria:

* Pregnancy
* Cardiac arrest of any cause as the indication for intubation
* Patient or next-of-kin declining participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be adult patients requiring emergent tracheal intubation for acute respiratory failure, coma, or shock, while cared for by an Emergency Physician either in the prehospital setting or in the hospital Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
number of missing items of the MACOCHA score | 5 minutes
  The MACOCHA score is a predictive score of difficult intubation in intensive care to anticipate and prepare the appropriate equipment, possibly use an alternative strategy of intubation and call for help to reduce the risk of morbidity and mortality.
  The MACOCHA score involves various simple assessment items: a Mallampati III or IV, a sleep apnea syndrome, a decrease in cervical mobility, a mouth opening <3cm, a coma defined by a Glasgow score <8, severe hypoxemia, and if the practitioner is not anesthetist.
  Missing items are defined as those for which relevant information cannot be collected before intubation.

SECONDARY OUTCOMES:
Adverse events | 30 min
  occurrence of any adverse event during and 30 minutes after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh Nay, MD, Principal Investigator — Centre Hospitalier régional d'Orléans, Orléans, France
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Jong A, Molinari N, Terzi N, Mongardon N, Arnal JM, Guitton C, Allaouchiche B, Paugam-Burtz C, Constantin JM, Lefrant JY, Leone M, Papazian L, Asehnoune K, Maziers N, Azoulay E, Pradel G, Jung B, Jaber S; AzuRea Network for the Frida-Rea Study Group. Early identification of patients at risk for difficult intubation in the intensive care unit: development and validation of the MACOCHA score in a multicenter cohort study. Am J Respir Crit Care Med. 2013 Apr 15;187(8):832-9. doi: 10.1164/rccm.201210-1851OC. PMID 23348979